CLINICAL TRIAL: NCT05478161
Title: Investigation of the Safety and Performance of the NVT ALLEGRA THV System With a New Delivery System in Patients With Severe Calcified Aortic Stenosis or Failed Surgical Aortic Bioprosthesis
Brief Title: Investigation of the ALLEGRA THV System With a New Delivery System in Patients With Aortic Stenosis or Failed Surgical Bioprosthesis
Acronym: EMPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NVT GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVT05EMP
Record Dates: First submitted 2022-07-19; First posted 2022-07-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Transcatheter Aortic Valve Implantation
Keywords: TAVI; Aortic valve stenosis; ALLEGRA; IMPERIA
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): TAVI in severe calcified aortic stenosis or in failed surgical aortic bioprosthesis
  Interventions: Device: (ALLEGRA Transcatheter Heart Valve) TAVI in severe calcified aortic stenosis or in failed surgical aortic bioprosthesis

INTERVENTIONS:
Device: (ALLEGRA Transcatheter Heart Valve) TAVI in severe calcified aortic stenosis or in failed surgical aortic bioprosthesis — Implantation of the ALLEGRA Transcatheter Heart Valve in failing surgical bioprosthesis

SUMMARY:
The EMPIRE study confirms the technical performance of the new IMPERIA Delivery System and evaluates the safety and efficacy of the entire ALLEGRA THV System.

The primary endpoint is device success rate at 7 days (discharge from index procedure or 7 days post implant, whichever comes first), as defined by VARC 2.

Based on the outcomes of a study with a similar device and considering a drop-out rate of 5%, 107 patients need to be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic severe calcific stenosis of a native aortic valve with an AVA ≤1.0 cm2 (or AVA index ≤0.6 cm2/m2), AND mean aortic pressure gradient ≥ 40mmHg OR maximal transaortic velocity ≥4.0m/s OR Doppler velocity index ≤0.25 on site-reported echocardiography OR symptomatic patients with degeneration of a surgical bioprosthetic valve (stenosis +/- insufficiency) on site-reported echocardiography
2. Local multi-disciplinary Heart Team and Central Screening Committee (CSC) agree on indication and eligibility for TAVI
3. Age ≥18 years
4. Patient has signed the Patient Informed Consent Form
5. Patient is willing and able to comply with requirements of the study, including all follow-up visits

Exclusion Criteria:

General:

1. Mean aortic annulus diameter as measured by pre-procedural CT or internal diameter of the bioprosthesis is <16.5 mm or >27 mm
2. Echocardiographic evidence of intracardiac thrombus or vegetation (site-reported)
3. Significant disease of the aorta that would preclude safe advancement of the ALLEGRA THV System
4. Severe ilio-femoral vessel disease that would preclude safe placement of an 18 Fr introducer sheath or make endovascular access impossible
5. Porcelain aorta
6. Severe left ventricular dysfunction with ejection fraction (EF) <20% (site-reported)
7. Evidence of active endocarditis or other acute infections
8. Renal failure requiring continuous renal replacement therapy
9. Untreated clinically significant coronary artery disease requiring revascularization
10. Any percutaneous interventional procedure (e.g. PCI with stenting) within 14 days prior of the index procedure
11. Acute MI ≤30 days prior to the index procedure
12. Symptomatic carotid or vertebral artery disease requiring intervention or carotid/vertebral intervention within the preceding 45 days
13. Cerebrovascular accident (CVA) or transient ischemic attack (TIA) ≤6 months or prior CVA with moderate or severe disability (e.g. modified Rankin scale score >2)
14. History of bleeding diathesis or coagulopathy; acute blood dyscrasias as defined: thrombocytopenia (platelets <80,000/µl), acute anemia (hemoglobin <10 g/dl), leukopenia (WBC <3000/ µl)
15. Active peptic ulcer or gastrointestinal (GI) bleeding ≤3 months
16. Severe (greater than 3+) mitral insufficiency (site-reported)
17. Uncontrolled atrial fibrillation
18. Required emergency surgery for any reason
19. Known hypersensitivity to contrast media, which cannot be adequately pre-medicated or contraindication to anticoagulant or anti-platelet medication or to nitinol alloy or to bovine tissue
20. Life expectancy ≤12 months due to other medical illness
21. Currently participating in another investigational drug or device study
22. Pregnancy or intend to become pregnant during study participation

    Specific exclusions in patients with native aortic valve disease (site-reported):
23. Unicuspid or bicuspid aortic valve
24. Non-calcified aortic stenosis
25. Predominant aortic regurgitation > grade 3
26. Distance between native aortic valve basal plane and the orifice of the lowest coronary artery <8 mm

    Specific exclusions in patients with degenerated surgical bioprosthetic aortic valves (valve-in-valve) (site-reported):
27. Low position of the coronary ostia, especially in combination with shallow sinuses (high risk of coronary occlusion)
28. Partially detached leaflets that may obstruct a coronary ostium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Device success at 7 days | 7 day
  * Absence of procedural mortality AND
  * Correct positioning of a single device in the proper anatomical location (site-reported) AND
  * Intended performance of the prosthetic heart valve (as determined by an independent Echo Core Lab at discharge from index procedure or 7 days post implant, whichever comes first)
    * Indexed Effective Orifice Area (iEOA) > 0.85 cm2/m2 for BMI < 30kg/m2 and iEOA > 0.70 cm2/m2 for BMI ≥ 30kg/m2
    * Mean aortic valve gradient <20 mmHg or peak velocity <3 m/s
    * No moderate or severe prosthetic valve regurgitation

SECONDARY OUTCOMES:
All-cause mortality | up to 12 months
Cardiovascular mortality | up to 12 months
All stroke | up to 12 months
TIA | up to 12 months
Procedural success | assessed immediately after the procedure
  * Successful vascular access, delivery and deployment of the ALLEGRA THV including re- positioning if required and successful retrieval of the IMPERIA Delivery System (site- reported)
  * Correct position of the ALLEGRA THV (site-reported)
  * Only one ALLEGRA THV implanted in proper anatomical position (site-reported)
Effective orifice area (EOA) as assessed by transthoracic echocardiogram (TTE) | up to 12 months
Transvalvular mean and peak pressure gradient as assessed by transthoracic echocardiogram (TTE) | up to 12 months
Trans- and paravalvular regurgitation as assessed by transthoracic echocardiogram (TTE) | up to 12 months
NYHA classification | 30 days, 6 months, and 12 months
Early safety | up to 30 days
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury-Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure (BAV, TAVI, or SAVR)
Time-related valve safety | up to 12 months
  * Structural valve deterioration
  * Valve-related dysfunction (mean aortic valve gradient
    * 20 mmHg, EOA ≤0.9-1.1 cm2c and/or DVI <0.35 m/s, AND/OR moderate or severe prosthetic valve regurgitation)
  * Requiring repeat procedure (TAVI or SAVR)
  * Prosthetic valve endocarditis
  * Prosthetic valve thrombosis
  * Thrombo-embolic events (e.g. stroke)
  * VARC bleeding, unless clearly unrelated to valve therapy (e.g. trauma)
Quality of life as assessed using the Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | up to 12 months
  Assessed with the Kansas City Cardiomyopathy Questionnaire (KCCQ-12). Patients are asked questions about physical limitation, symptom frequency, quality of life, and social limitation. Responses are given on a Likert scale that for each individual item is scored on a scale of 0-100 with higher scores indicating better health.
New pacemaker implantation | up to 12 months
Delivery system related AEs | discharge from index procedure or 7 days post implant, whichever comes first

CONTACTS AND LOCATIONS:
Locations (2):
- Schüchtermann Klinik, Bad Rothenfelde, Lower Saxony, Germany
- Hospital Alvaro Cunqueiro, Vigo, Spain